CLINICAL TRIAL: NCT06818721
Title: Intravitreal Topotecan for the Prevention or Treatment of Proliferative Vitreoretinopathy in Patients with Rhegmatogenous Retinal Detachment: a Prospective Matched Cohort Study
Brief Title: Intravitreal Topotecan for Prevention or Treatment of Proliferative Vitreoretinopathy in Retinal Detachment
Acronym: TOPO-PT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOPO-PT
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Retinal Detachment Rhegmatogenous; Proliferative Vitreoretinopathy
Keywords: topotecan; proliferative vitreoretinopathy; rhegmatogenous retinal detachment
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Topotecan; Scleral Buckling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravitreal topotecan with retinal detachment surgery (Experimental): Intravitreal topotecan 8 µg/0.05mL, diluted in sterile saline and administered preoperatively, within one week prior to surgery, as well as one week postoperatively.
  Interventions: Drug: Intravitreal topotecan; Procedure: Retinal detachment surgery
- Retinal detachment surgery (Active Comparator): Historical control patients who previously received standard of care surgery for rhegmatogenous retinal detachment without intravitreal topotecan.
  Interventions: Procedure: Retinal detachment surgery

INTERVENTIONS:
Drug: Intravitreal topotecan — Patients who meet all inclusion criteria and none of the exclusion criteria will receive intravitreal topotecan (8 µg in 0.05 mL). The treatment will be administered within one week before retinal detachment surgery (pneumatic retinopexy, pars plana vitrectomy, and/or scleral buckling) and one week after surgery, for a total of two injections.
  Other Names: Topotecan
  Arms: Intravitreal topotecan with retinal detachment surgery
Procedure: Retinal detachment surgery — Standard retinal detachment surgery (pneumatic retinopexy, three-port pars plana vitrectomy, and/or scleral buckling).
  Other Names: Pars plana vitrectomy; Pneumatic retinopexy; Scleral buckling

SUMMARY:
Intravitreal topotecan exhibits strong anti-inflammatory, anti-proliferative, and anti-fibrotic properties, making it a promising option for preventing and treating proliferative vitreoretinopathy in rhegmatogenous retinal detachment. Preclinical studies have demonstrated its efficacy in proliferative vitreoretinopathy models, where no adverse events have been reported for doses of 5 µg to 30 µg. This prospective, matched cohort study aims to assess the therapeutic efficacy and safety of intravitreal topotecan for preventing and treating proliferative vitreoretinopathy in rhegmatogenous retinal detachment patients.

DETAILED DESCRIPTION:
Patients who provide informed consent for participation in the experimental study arm will undergo standard-of-care retinal detachment surgery with intravitreal topotecan (8 µg/0.05 mL), diluted in sterile saline and administered preoperatively within one week before surgery, as well as one week postoperatively. Matched historical control patients who received standard-of-care retinal detachment surgery without intravitreal topotecan will be eligible for study participation. Both the experimental and historical control study arms will be further divided into two groups: (i) patients with rhegmatogenous retinal detachment who exhibit high-risk characteristics of proliferative vitreoretinopathy on optical coherence tomography or have early proliferative vitreoretinopathy confirmed by clinical examination, and (ii) patients with rhegmatogenous retinal detachment who have neither high-risk characteristics of proliferative vitreoretinopathy nor a history of proliferative vitreoretinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and older
2. Patients who undergo pneumatic retinopexy, pars plana vitrectomy and/or scleral buckling for rhegmatogenous retinal detachment
3. Patients who are voluntarily able and willing to participate

Patients undergoing combined phacoemulsification and pars plana vitrectomy and/or scleral buckling will also be included. Any surgical technique will be considered, including relaxing retinotomy or retinectomy during pars plana vitrectomy.

Exclusion Criteria:

1. Patients with a history of exudative retinal detachment
2. Patients with severe non-proliferative or proliferative diabetic retinopathy
3. Patients with other planned ocular surgery following pars plana vitrectomy
4. Female patients of childbearing age (i.e. less than 50 years old) who intend to become pregnant over the course of the study
5. Patients with pre-existing bone marrow suppression or cytopenias
6. Patients with pre-existing interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrent rhegmatogenous retinal detachment secondary to proliferative vitreoretinopathy | 6 months or last follow-up

SECONDARY OUTCOMES:
Grade of proliferative vitreoretinopathy | 6 months or last follow-up
Rate of primary retinal reattachment | 6 months or last follow-up
Rate of final retinal reattachment | 6 months or last follow-up
Best-corrected visual acuity | 6 months or last follow-up
Change in best-corrected visual acuity from baseline | 6 months or last follow-up
Rate of complications | 6 months or last follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No